CLINICAL TRIAL: NCT00432861
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Crossover Study to Evaluate the Effectiveness and Safety of PANCRECARB® MS-16 (Pancrelipase) in Reducing Steatorrhea in Children and Adults With Cystic Fibrosis
Brief Title: Evaluation of the Safety and Efficacy of Pancrecarb® MS-16 in Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Digestive Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pancrecarb; DCI 06-001
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Cystic Fibrosis; Pancreatic Insufficiency
Keywords: cystic fibrosis; pancreatic insufficiency; PANCRECARB® MS-16 (pancrelipase); steatorrhea
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Steatorrhea | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pancrecarb(R) MS-16 Capsules
  Interventions: Drug: PANCRECARB® (pancrelipase)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PANCRECARB® (pancrelipase) — Capsules
  Other Names: MS-16
  Arms: 1
Drug: Placebo — Capsules
  Arms: 2

SUMMARY:
The primary objective of this study is to determine if PANCRECARB® MS-16 (pancrelipase) is safe and effective in reducing steatorrhea (as measured by 72-hour stool fat determinations) in children and adults with cystic fibrosis and pancreatic insufficiency.

DETAILED DESCRIPTION:
Pancreatic insufficiency (PI) is a common pathologic condition that occurs in approximately 90% of patients with cystic fibrosis (CF). Pancreatic insufficiency is characterized by both pancreatic enzyme and bicarbonate insufficiencies. Consequently, maldigestion occurs and a variety of essential nutrients are lost through the stools, especially fat and fat soluble vitamins. As a result, patients often experience growth failure and malnutrition. Effective correction of maldigestion is critical to the survival and well-being of these patients.

Several strengths of PANCRECARB® (pancrelipase) (i.e., MS4, MS8, MS16) have been available and used by patients with CF for more than a decade. The digestive enzymes in PANCRECARB® (pancrelipase) act locally in the gastrointestinal tract. The active enzymes hydrolyze fats into glycerol and fatty acids, proteins into peptides and amino acids, and starches into dextrins and maltose. PANCRECARB® (pancrelipase) has the potential to promote increased lipase activity with efficient fat digestion. Efficient fat digestion is important in CF because it may lead to improved nutritional and pulmonary status and ultimately to improved quality of life and enhanced survival.

PANCRECARB® MS-8 (pancrelipase) has been compared to enteric-coated pancreatic enzymes without bicarbonate for its efficacy in reducing steatorrhea in patients with CF. Differences in fat excretion, when subjects received PANCRECARB® MS-8 (pancrelipase) versus enteric-coated enzymes without bicarbonate, were compared using linear modeling. Mean fat excretion decreased significantly in subjects who received PANCRECARB® MS-8 (pancrelipase) compared to enteric-coated enzymes without bicarbonate.

This study has been designed in accordance with FDA 2006 guideline on exocrine pancreatic insufficiency drug products. Assuming that the results of this study demonstrate that therapy with PANCRECARB® MS-16 (pancrelipase) results in clinically and statistically significant improvement in fat absorption relative to placebo in subjects with CF and pancreatic insufficiency, the study results will be part of a submission for marketing approval of PANCRECARB® (pancrelipase).

The study consists of two treatment periods with 72-hour stool collections separated by a washout period. Study subjects will be required to consume a diet high in fat content.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 7 years
* Confirmed diagnosis of CF based on the following criteria: One or more clinical features consistent with the CF phenotype, AND Positive sweat chloride ≥ 60 mEq/liter (by pilocarpine iontophoresis), OR Genotype with two identifiable mutations consistent with CF
* Adequate nutritional status based on BMI: Age 7 years to 20 years old, Body Mass Index Percentile ≥ 5th percentile; Age > 20 years old, Body Mass Index for females ≥ 16.0, Body Mass Index for males ≥ 16.5
* Pancreatic insufficiency documented by spot fecal elastase-1 (FE 1) <= 100 micrograms/g stool at the time of randomization
* Currently receiving pancreatic enzyme replacement therapy with a commercially available pancreatic enzyme
* Able to swallow size 0 capsules
* Clinically stable with no evidence of an acute medical condition
* Able to understand and sign a written informed consent or assent and comply with the requirements of the study

Exclusion Criteria:

* History of fibrosing colonopathy
* History of significant bowel resection
* History of being refractory to pancreatic enzyme replacement therapy
* Solid organ transplant
* Abdominal surgery within past five (5) years
* A current diagnosis or a history of distal intestinal obstruction syndrome (DIOS) in the past six (6) months, or 2 or more episodes of DIOS in the past twelve (12) months
* Conditions known to increase fecal fat loss including: inflammatory bowel disease , celiac disease, Crohn's disease, tropical Sprue, Whipple's disease
* A known contraindication, sensitivity or hypersensitivity to porcine pancreatic enzymes or food dyes (i.e., FD&C Blue No. 2)
* Active liver disease with liver enzymes (alanine aminotransferase (ALT/SGPT), aspartate aminotransferase (AST/SGOT) or bilirubin ≥ 3 times the upper limit of normal
* Acute pancreatitis or acute exacerbation of chronic pancreatitis
* Acute treatment with any systemic (oral or IV) antibiotics two (2) weeks prior to screening
* Treatment with erythromycin and unwilling to discontinue the treatment two (2) weeks prior to the screening. (azithromycin is allowed)
* Change in chronic treatment with systemic (oral and IV) antibiotics during the trial NOTE: Study subject may remain on a chronic regimen of systemic (oral or IV) antibiotics (with exception of erythromycin), if he/she started the antibiotics at least 2 weeks prior to study screening, was at his/her usual bowel pattern at the time of screening, and does not stop or change these antibiotics during the study period.
* Receiving enteral tube feeding during the study
* Expected inability to cooperate with or be non-adherent to required study procedures
* Pregnant, breast-feeding, or unwilling to practice birth control (for females of child-bearing potential) during participation in the study
* Use of narcotics
* Poorly controlled diabetes
* Participation in an investigational study of a drug, biologic, or device not currently approved for marketing, within 30 days of screening visit
* A medical condition which the investigator deems significant enough to interfere with the ability of the study patient to participate in the trial or interfering with assessment of effects of enzyme therapy on fat absorption

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
percent coefficient of fat absorption (% CFA) | calculated from the 72-hour stool collection and dietary records

SECONDARY OUTCOMES:
percent coefficient of nitrogen absorption (% CNA) | calculated from the 72-hour stool collections and dietary records
change in stool frequency and stool weight | recorded over the 72-hour stool collection period

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Konstan, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

REFERENCES:
- [Background] Davis PB, Drumm M, Konstan MW. Cystic fibrosis. Am J Respir Crit Care Med. 1996 Nov;154(5):1229-56. doi: 10.1164/ajrccm.154.5.8912731. No abstract available.
- [Background] Borowitz D, Baker RD, Stallings V. Consensus report on nutrition for pediatric patients with cystic fibrosis. J Pediatr Gastroenterol Nutr. 2002 Sep;35(3):246-59. doi: 10.1097/00005176-200209000-00004. No abstract available. PMID 12352509
- [Background] Brady MS, Garson JL, Krug SK, Kaul A, Rickard KA, Caffrey HH, Fineberg N, Balistreri WF, Stevens JC. An enteric-coated high-buffered pancrelipase reduces steatorrhea in patients with cystic fibrosis: a prospective, randomized study. J Am Diet Assoc. 2006 Aug;106(8):1181-6. doi: 10.1016/j.jada.2006.05.011. PMID 16863712
- [Background] Borowitz DS, Grand RJ, Durie PR. Use of pancreatic enzyme supplements for patients with cystic fibrosis in the context of fibrosing colonopathy. Consensus Committee. J Pediatr. 1995 Nov;127(5):681-4. doi: 10.1016/s0022-3476(95)70153-2. No abstract available. PMID 7472816
- [Background] Konstan MW, Stern RC, Trout JR, Sherman JM, Eigen H, Wagener JS, Duggan C, Wohl ME, Colin P. Ultrase MT12 and Ultrase MT20 in the treatment of exocrine pancreatic insufficiency in cystic fibrosis: safety and efficacy. Aliment Pharmacol Ther. 2004 Dec;20(11-12):1365-71. doi: 10.1111/j.1365-2036.2004.02261.x. PMID 15606399
- [Background] Rosenstein BJ, Cutting GR. The diagnosis of cystic fibrosis: a consensus statement. Cystic Fibrosis Foundation Consensus Panel. J Pediatr. 1998 Apr;132(4):589-95. doi: 10.1016/s0022-3476(98)70344-0. PMID 9580754
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Borowitz D, Baker SS, Duffy L, Baker RD, Fitzpatrick L, Gyamfi J, Jarembek K. Use of fecal elastase-1 to classify pancreatic status in patients with cystic fibrosis. J Pediatr. 2004 Sep;145(3):322-6. doi: 10.1016/j.jpeds.2004.04.049. PMID 15343184
- [Background] Stern RC, Eisenberg JD, Wagener JS, Ahrens R, Rock M, doPico G, Orenstein DM. A comparison of the efficacy and tolerance of pancrelipase and placebo in the treatment of steatorrhea in cystic fibrosis patients with clinical exocrine pancreatic insufficiency. Am J Gastroenterol. 2000 Aug;95(8):1932-8. doi: 10.1111/j.1572-0241.2000.02244.x. PMID 10950038
- [Background] VAN DE KAMER JH, TEN BOKKEL HUININK H, WEYERS HA. Rapid method for the determination of fat in feces. J Biol Chem. 1949 Jan;177(1):347-55. No abstract available. PMID 18107439
- See also: Digestive Care, Inc. — http://www.digestivecare.com